CLINICAL TRIAL: NCT00715403
Title: Extension Study to Establish Safety, Pharmacokinetics and Efficacy of BIBF 1120 in Patients With Previous Clinical Benefit From BIBF 1120
Brief Title: A Phase I/II Open Label Extension Study of BIBF 1120 Administered Orally Once or Twice Daily to Establish Safety, Pharmacokinetics and Efficacy in Patients With Advanced Solid Tumours and Clinical Benefit From Previous Therapy With BIBF 1120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1199.16
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — nintedanib

INTERVENTIONS:
Drug: BIBF 1120

SUMMARY:
The primary objective of this trial is to evaluate the long-term safety of BIBF 1120 in terms of incidence and intensity of Adverse Events and changes in safety laboratory parameters.

Secondary objectives are the collection of further safety data (vital signs), efficacy data and the determination of pharmacokinetic characteristics during long-term therapy with BIBF 1120.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with advanced solid tumours who have completed a previous study with BIBF 1120. The patients should not have progression of their underlying tumour disease unless there is evidence for significant clinical benefit (e.g. symptom improvement) from treatment with BIBF 1120.
2. Age 18 years or older
3. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score <= 2
4. Patients must have given written informed consent (which must be consistent with ICH-GCP and local legislation)

Exclusion Criteria:

1. Time elapsed from last administration of BIBF 1120 in the previous trial to start of treatment in the present trial exceeds four weeks
2. Presence of drug related toxicity > grade 2 CTC from previous therapy with BIBF 1120 or presence of drug related continuous toxicity of grade 2 for seven or more consecutive days which would preclude ongoing chronic therapy with BIBF 1120
3. Active ulcers (gastro-intestinal tract, skin)
4. Major injuries and surgery within the past three weeks with incomplete wound healing
5. Hypersensitivity to BIBF 1120 or the excipients of the trial drug
6. Known secondary malignancy requiring therapy
7. Active infectious disease
8. Significant cardiovascular diseases (i.e. uncontrolled severe hypertension, unstable angina pectoris, history of myocardial infarction, congestive heart failure > NYHA II)
9. Gastrointestinal disorders anticipated to interfere with the resorption of the study drug
10. Brain metastases requiring therapy
11. Absolute neutrophil count less than 1,500/mm3
12. Platelet count less than 100,000/mm3
13. Bilirubin greater than 1.5 mg/dl (> 26 µmol/L)
14. Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
15. Serum creatinine greater than 2 mg/dl (> 176 µmol/L)
16. Concomitant non-oncological diseases which are considered relevant for the evaluation of the safety of the trial drug
17. Chemo-, radio-, or immunotherapy within the past four weeks prior to treatment with the trial drug
18. Patients who are sexually active and unwilling to use a medically acceptable method of contraception
19. Pregnancy or lactation
20. Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy (visit 2) or concomitantly with this trial (except for a previous study with BIBF 1120)
21. Patients unable to comply with the protocol
22. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- France (7):
  - 1199.16.3306A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1199.16.3311A Boehringer Ingelheim Investigational Site, Clichy
  - 1199.16.3311B Boehringer Ingelheim Investigational Site, Clichy
  - 1199.16.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1199.16.3312A Boehringer Ingelheim Investigational Site, Paris
  - 1199.16.3313A Boehringer Ingelheim Investigational Site, Paris
  - 1199.16.3313E Boehringer Ingelheim Investigational Site, Paris
- Germany (4):
  - 1199.16.49001 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1199.16.49004 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1199.16.49008 Boehringer Ingelheim Investigational Site, Tübingen
  - 1199.16.49005 Boehringer Ingelheim Investigational Site, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multinational, open-label, uncontrolled, extension trial with Nintedanib in patients who had experienced a clinical benefit with Nintedanib (objective tumour response or disease stabilisation and/or symptom improvement) in either one out of five phase I or phase I/IIA clinical trials for advanced solid tumours at study entry.
Groups:
- 50mg QD: Patients were treated with 50 mg Nintedanib once daily (QD) in the morning.
- 200mg QD: Patients were treated with 200 mg Nintedanib once daily in the morning.
- 100mg BID: Patients were treated with 100 mg Nintedanib twice daily (BID).
- 150mg BID: Patients were treated with 150 mg Nintedanib twice daily.
- 200mg BID: Patients were treated with 200 mg Nintedanib twice daily.
- 250mg BID: Patients were treated with 250 mg Nintedanib twice daily.
- 300mg BID: Patients were treated with 300 mg Nintedanib twice daily.
Period: Overall Study
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Started | 1 | 1 | 4 | 9 | 6 | 19 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 4 | 9 | 6 | 19 | 1
Not completed — Progressive disease | 0 | 1 | 3 | 9 | 5 | 14 | 1
Not completed — Dose limiting Toxicity (DLT) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Adverse Event than DLT | 1 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reason not defined above | 0 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which comprised of all patients who received at least one dose of Nintedanib in both their previous Nintedanib trial and in this extension trial
Groups:
- 50mg QD: Patients were treated with 50 mg Nintedanib once daily in the morning.
- 100mg BID: Patients were treated with 100 mg Nintedanib twice daily.
- Total: Total of all reporting groups
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID | Total
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1 | 41
Age, Continuous [Median (Full Range); unit: years] | 75.0 [75 to 75] | 47.0 [47 to 47] | 65.5 [52 to 75] | 66.0 [52 to 78] | 63.5 [45 to 74] | 66.0 [41 to 80] | 67.0 [67 to 67] | 66.0 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 8
  Male | 1 | 0 | 2 | 7 | 4 | 18 | 1 | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Intensity of Adverse Events With Highest CTCAE Grade 1
Description: All patients who had grade 1 adverse events (AEs) as the worst grade of the AE. Incidence and intensity of Adverse Events with grading of Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From signing the informed consent until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Dyspepsia | 100 | 0 | 0 | 11 | 0 | 0 | 0
  Fatigue | 100 | 0 | 0 | 33 | 17 | 0 | 0
  Nasopharyngitis | 100 | 0 | 0 | 0 | 33 | 5 | 0
  Anorexia | 100 | 0 | 0 | 11 | 0 | 16 | 0
  Hyperhidrosis | 100 | 0 | 0 | 11 | 0 | 5 | 0
  Diarrhoea | 0 | 100 | 0 | 44 | 50 | 37 | 100
  Bronchitis | 0 | 100 | 0 | 0 | 0 | 0 | 0
  Eye disorder | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Eyelid oedema | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Haemorrhoids | 0 | 0 | 25 | 0 | 0 | 5 | 0
  Toothache | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 0 | 25 | 11 | 17 | 5 | 0
  Muscle spasms | 0 | 0 | 25 | 11 | 0 | 11 | 0
  Neck pain | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Pain in extremity | 0 | 0 | 25 | 11 | 17 | 5 | 0
  Vulvovaginal dryness | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Arrhythmia | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 33 | 67 | 21 | 0
  Vomiting | 0 | 0 | 0 | 22 | 33 | 5 | 0
  Abdominal pain | 0 | 0 | 0 | 11 | 33 | 11 | 0
  Gastrooesophageal reflux disease | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Tooth discolouration | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Asthenia | 0 | 0 | 0 | 11 | 33 | 5 | 0
  Xerosis | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Gastrointestinal infection | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Bone pain | 0 | 0 | 0 | 22 | 17 | 0 | 0
  Arthralgia | 0 | 0 | 0 | 11 | 50 | 5 | 0
  Musculoskeletal chest pain | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Myalgia | 0 | 0 | 0 | 11 | 0 | 0 | 100
  Dizziness | 0 | 0 | 0 | 22 | 0 | 5 | 0
  Headache | 0 | 0 | 0 | 11 | 0 | 5 | 0
  Anxiety | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Rales | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Nail disorder | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Hot flush | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Vertigo | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 17 | 16 | 0
  Flatulence | 0 | 0 | 0 | 0 | 17 | 11 | 0
  Gastric disorder | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Hypersensitivity | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Viral infection | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Musculoskeletal pain | 0 | 0 | 0 | 0 | 17 | 5 | 0
  Balance disorder | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Carpal tunnel syndrome | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Sciatica | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Dysuria | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 0 | 33 | 0 | 0
  Rash maculo-papular | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Eye pain | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Visual impairment | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Abdominal distension | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Gastrointestinal haemorrhage | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Adverse drug reaction | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Chest pain | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Chills | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Hepatic pain | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Urinary tract infection | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Weight decreased | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Hyperglycaemia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Muscular weakness | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Back pain | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Joint swelling | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Dysgeusia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Peripheral sensory neuropathy | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Insomnia | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Haematuria | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Incontinence | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Alopecia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Dry skin | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Pruritus | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Conjunctivitis | 0 | 0 | 0 | 0 | 0 | 0 | 100
  Haemoptysis | 0 | 0 | 0 | 0 | 0 | 0 | 100

2. Secondary Outcome: Clinically Relevant Abnormalities for Vital Signs
Description: Clinically relevant abnormalities for Vital Signs (systolic blood pressure, diastolic blood pressure, and pulse rate). New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: From baseline until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Pre-dose Concentration of Nintedanib in Plasma at Steady-state (Cpre,ss)
Description: Cpre,ss represents the pre-dose concentration of Nintedanib in Plasma at steady-state at day 29
Time Frame: Just before drug administration every 28±7 days after day 29
Population: Treated set. No descriptive statistics could be calculated for the dosing groups 50 mg and 200 mg QD; 100 mg and 300 mg BID due to insufficient patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 2 | 7 | 0
ng/mL |  |  |  | 7.54 (48.3) | 11.8 (33.5) | 11.0 (48.5) |

4. Secondary Outcome: Unconfirmed Best Overall Response
Description: Unconfirmed best overall response assessed by RECIST (Response Evaluation Criteria In Solid Tumours) criteria (version 1.0).
  PD = Progressive disease.
Time Frame: Baseline until end of treatment, up to 991 days
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Complete response | 0 | 100 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Stable disease | 100 | 0 | 75 | 33 | 0 | 16 | 0
  Non-evaluable, clinically non-progressive disease | 0 | 0 | 25 | 11 | 83 | 5 | 0
  PD or non-evaluable , clinically PD | 0 | 0 | 0 | 11 | 17 | 32 | 100
  Unknown | 0 | 0 | 0 | 44 | 0 | 42 | 0

5. Secondary Outcome: Unconfirmed Best Objective Response
Description: Unconfirmed best objective response assessed by RECIST (Response Evaluation Criteria In Solid Tumours) criteria (version 1.0)
Time Frame: Baseline until end of treatment, up to 991 days
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  No | 100 | 0 | 100 | 56 | 100 | 53 | 100
  Yes | 0 | 100 | 0 | 0 | 0 | 5 | 0
  Unknown | 0 | 0 | 0 | 44 | 0 | 42 | 0

6. Secondary Outcome: Clinical Benefit
Description: Clinical benefit was defined as the absence of disease progression (no PD or nonevaluable clinically progressive disease) determined by RECIST (version 1.0).
Time Frame: Baseline until end of treatment, up to 991 days
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  No | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Yes | 100 | 100 | 100 | 100 | 100 | 89 | 100

7. Secondary Outcome: Confirmed Objective Response
Description: Confirmed objective response assessed by RECIST (Response Evaluation Criteria In Solid Tumours) criteria (version 1.0)
Time Frame: Baseline until end of treatment, up to 991 days
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  No | 100 | 0 | 100 | 56 | 100 | 58 | 100
  Yes | 0 | 100 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 44 | 0 | 42 | 0

8. Secondary Outcome: Progression Free Survival
Description: Percentage of participants that experienced progression free survival (PFS), assessed by RECIST (Response Evaluation Criteria In Solid Tumours) (version 1.0), by day 1230. Progression was defined as progressive disease (PD) or non-evaluable clinically progressive disease.
  PFS was defined for patients without PD at screening as the time from first treatment with the trial drug in the previous trial until onset of PD or death, whatever comes earlier.
  Patients with PD could enter the trial if they showed signs of clinical benefit. For patients with PD at screening, the RECIST assessment at screening was used as a new baseline value and PFS was the time from first treatment with the trial drug in this trial until the onset of progressive disease in this trial or death, whatever comes first.
Time Frame: First drug administration (in previous trial) until end of treatment, up to 1230 days
Population: Treated set. Data for category
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Progression (RECIST) | 0 | 100 | 25 | 11 | 33 | 42 | 100
  Death | 0 | 0 | 0 | 0 | 0 | 32 | 0
  No progressive disease (RECIST) or death | 100 | 0 | 75 | 44 | 67 | 16 | 0
  Unknown | 0 | 0 | 0 | 45 | 0 | 10 | 0

9. Primary Outcome: Incidence and Intensity of Adverse Events With Highest CTCAE Grade 2
Description: All patients who had grade 2 adverse events (AEs) as the worst grade of the AE. Incidence and intensity of Adverse Events with grading of Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From signing the informed consent until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Fatigue | 0 | 0 | 0 | 22 | 0 | 11 | 0
  Anorexia | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Diarrhoea | 0 | 0 | 0 | 11 | 33 | 21 | 0
  Bronchitis | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Abdominal pain | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Asthenia | 0 | 0 | 25 | 11 | 0 | 11 | 0
  Gastrointestinal infection | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Bone pain | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Arthralgia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Musculoskeletal chest pain | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Headache | 0 | 0 | 25 | 11 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Flatulence | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Musculoskeletal pain | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Sciatica | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Dyspnoea | 0 | 0 | 0 | 11 | 0 | 11 | 0
  Chest pain | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Urinary tract infection | 0 | 0 | 25 | 0 | 0 | 5 | 0
  Weight decreased | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Back pain | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Peripheral sensory neuropathy | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Haemoptysis | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Osteoarthritis | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Parotitis | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Osteolysis | 0 | 0 | 0 | 11 | 0 | 0 | 0
  Abdominal pain upper | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Gastrointestinal disorder | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Groin pain | 0 | 0 | 0 | 0 | 17 | 0 | 0
  Anaemia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Oedema peripheral | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Dehydration | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Productive cough | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Deep vein thrombosis | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Phlebitis superficial | 0 | 0 | 0 | 0 | 0 | 5 | 0

10. Primary Outcome: Incidence and Intensity of Adverse Events With Highest CTCAE Grade 3
Description: All patients who had grade 3 adverse events (AEs) as the worst grade of the AE. Incidence and intensity of Adverse Events with grading of Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From signing the informed consent until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Gamma-glutamyltransferase increased | 100 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhoea | 0 | 0 | 25 | 11 | 0 | 5 | 0
  Diarrhoea infectious | 0 | 0 | 25 | 0 | 0 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 11 | 0 | 5 | 0
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Haemorrhoids | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Ileus | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Subileus | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Pneumonia | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Convulsion | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Renal failure | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Urinary tract obstruction | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Pleural effusion | 0 | 0 | 0 | 0 | 0 | 5 | 0

11. Primary Outcome: Incidence and Intensity of Adverse Events With Highest CTCAE Grade 4
Description: All patients who had grade 4 adverse events (AEs) as the worst grade of the AE. Incidence and intensity of Adverse Events with grading of Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From signing the informed consent until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Incidence and Intensity of Adverse Events With Highest CTCAE Grade 5
Description: All patients who had grade 5 adverse events (AEs) as the worst grade of the AE. Incidence and intensity of Adverse Events with grading of Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From signing the informed consent until final follow-up, up to 991 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
percentage of participants
  Subdural Haematoma | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Malignant neoplasm progression | 0 | 0 | 0 | 0 | 0 | 26 | 0

13. Primary Outcome: Difference From Baseline for Liver Enzymes
Description: Difference from baseline (normalized value). Baseline was defined as the value at the time point closest to but prior to very first administration of trial medication. The standard error is actually the Interquartile Range calculated as P75 minus P25.
Time Frame: From signing the informed consent until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: U/L
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 18 | 1
U/L
  Alkaline phosphatase | 127.0 (0.0) | 11.9 (0.0) | -39.0 (70.5) | -21.2 (96.4) | -11.7 (81.0) | 16.0 (180.9) | 7.2 (0.0)
  Aspartate aminotransferase | 14.3 (0.0) | 13.7 (0.0) | 9.6 (18.0) | 6.8 (9.1) | 4.3 (41.0) | 15.9 (35.1) | 7.6 (0.0)
  Alanine aminotransferase | 10.6 (0.0) | 6.6 (0.0) | 0.6 (11.1) | -1.6 (18.8) | 9.1 (45.4) | 17.0 (33.6) | 12.4 (0.0)

14. Primary Outcome: Difference From Baseline for Bilirubin, Creatinine and Glucose
Description: as for outcome 13
Time Frame: From signing the informed consent until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: mg/dL
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 18 | 1
mg/dL
  Bilirubin (total) | 0.5 (0.0) | 0.0 (0.0) | 0.0 (0.2) | 0.0 (0.3) | 0.1 (0.1) | 0.1 (0.3) | 0.0 (0.0)
  Creatinine | -0.1 (0.0) | -0.3 (0.0) | 0.0 (0.2) | -0.1 (0.0) | -0.1 (0.2) | -0.1 (0.3) | 0.0 (0.0)
  Glucose (N=1,1,3,9,4,14,1) | -60.0 (0.0) | -2.2 (0.0) | 28.9 (126.1) | -11.3 (75.1) | -76.5 (75.9) | -23.3 (52.2) | -40.0 (0.0)

15. Primary Outcome: Difference From Baseline for Haemoglobin
Description: Difference from baseline for Haemoglobin (normalized value). Baseline was defined as the value at the time point closest to but prior to very first administration of trial medication. The standard error is actually the Interquartile Range calculated as P75 minus P25.
Time Frame: From baseline until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: g/dL
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 18 | 1
g/dL | -1.8 (0.0) | 1.4 (0.0) | 0.4 (2.3) | 1.0 (1.3) | 1.2 (0.7) | -0.2 (2.1) | 1.1 (0.0)

16. Primary Outcome: Difference From Baseline for Haematology and Differentials Parameters
Description: as for outcome 13
Time Frame: From signing the informed consent until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: 10^9 /L
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 18 | 1
10^9 /L
  Platelets | 42.2 (0.0) | 11.1 (0.0) | 1.0 (83.7) | -2.5 (25.2) | -38.1 (39.9) | 11.2 (65.9) | -27.1 (0.0)
  White blood cell count | -1.1 (0.0) | -0.7 (0.0) | 0.2 (2.9) | -0.8 (2.6) | -0.1 (5.6) | 0.7 (2.9) | 0.0 (0.0)
  Lymphocytes (N=1,1,4,9,4,17,1) | -0.6 (0.0) | -0.4 (0.0) | -0.1 (2.0) | 1.0 (1.1) | 0.0 (1.6) | 0.6 (0.6) | 1.1 (0.0)
  Neutrophils (N=1,1,4,9,6,17,1) | -4.1 (0.0) | -4.7 (0.0) | 0.9 (3.7) | -1.0 (5.6) | -2.4 (10.0) | -0.5 (3.0) | -1.2 (0.0)

17. Primary Outcome: Difference From Baseline for Coagulation Parameters
Description: Difference from baseline (normalized value) in coagulation parameters Prothrombin time, international normalised ratio (PT-INR) and partial thromboplastin time. Baseline was defined as the value at the time point closest to but prior to very first administration of trial medication. The standard error is actually the Interquartile Range calculated as P75 minus P25.
Time Frame: From signing the informed consent until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: sec
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
sec
  PT-INR (N=1,1,3,7,5,14,1) | 0.1 (0.0) | 0.1 (0.0) | 0.3 (0.6) | 0.1 (0.1) | 0.2 (0.5) | -0.0 (0.1) | 0.1 (0.0)
  Partial thromboplastin time (N=1,1,3,9,4,14,1) | 0.7 (0.0) | 2.6 (0.0) | -3.6 (6.7) | 1.9 (4.3) | 1.9 (4.3) | 1.5 (4.7) | -2.9 (0.0)

18. Primary Outcome: Difference From Baseline for Electrolytes
Description: as for outcome 13
Time Frame: From signing the informed consent until end of treatment, up to 991 days
Population: Treated set.
Measure: Median (Standard Error); unit: mmol/L
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Number analyzed (Participants) | 1 | 1 | 4 | 9 | 6 | 19 | 1
mmol/L
  Potassium (N=1,1,4,9,6,18,1) | 0.2 (0.0) | -0.3 (0.0) | -0.3 (2.1) | 0.1 (0.4) | -0.0 (1.1) | 0.1 (0.9) | 0.0 (0.0)
  Sodium (N=1,1,4,9,6,18,1) | 2.0 (0.0) | 1.0 (0.0) | 3.3 (5.2) | 0.0 (1.5) | 1.5 (6.0) | -1.3 (5.5) | 5.0 (0.0)

ADVERSE EVENTS:
Time Frame: From the first intake of trial medication until 28 days after last intake of medication, up to 1119 days
Arm/Group | 50mg QD | 200mg QD | 100mg BID | 150mg BID | 200mg BID | 250mg BID | 300mg BID
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 1/9 | 0/6 | 9/19 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 9/9 | 6/6 | 17/19 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50mg QD (N=1) | 200mg QD (N=1) | 100mg BID (N=4) | 150mg BID (N=9) | 200mg BID (N=6) | 250mg BID (N=19) | 300mg BID (N=1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50mg QD (N=1) | 200mg QD (N=1) | 100mg BID (N=4) | 150mg BID (N=9) | 200mg BID (N=6) | 250mg BID (N=19) | 300mg BID (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 6 | 5 | 12 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 4 | 6 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 2 | 3 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 5 | 1 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.